CLINICAL TRIAL: NCT03462134
Title: Can Orthopaedic Surgeons Predict the Outcome of Treatment in Patients With Meniscal Tears? The Results of an International Survey.
Brief Title: Predicting the Outcome After Treatment of Meniscal Tears
Status: Completed | Type: Observational
Sponsor: Onze Lieve Vrouwe Gasthuis (Other)
Collaborators: University of New South Wales (Unknown); Mayo Clinic (Other)
Responsible Party: Principal Investigator, Victor van de Graaf, principal investigator, Onze Lieve Vrouwe Gasthuis
Other Study IDs: 1
Record Dates: First submitted 2018-03-02; First posted 2018-03-12 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Meniscus Lesion; Surveys and Questionnaires
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Survey amongst orthopaedic surgeons: Selected of 20 patients from the Escape trial (NCT01850719)
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Survey amongst orthopaedic surgeons

SUMMARY:
In this study the investigators examined the ability of orthopaedic surgeons to predict the outcome of surgery and non-operative treatment in patients (age 45 to 70) with a non-obstructive meniscal tear.

DETAILED DESCRIPTION:
The additional benefits of Arthroscopic Partial Meniscectomy (APM) in middle aged patients with a non-obstructive meniscal tear are under scrutiny for years. Despite the most recent publications recommending to apply non-operative treatment (exercise therapy, injections, drugs) instead of APM in this patient group, the expected decrease in number of operations is slower then expected. Orthopaedic surgeons therefore seem unconvinced by the evidence to change practice.

For this reason the investigators conducted an international survey amongst orthopaedic surgeons in which the investigators aimed to (1) determine the ability of orthopaedic surgeons to predict the outcomes of APM and physical therapy (PT) in middle aged patients with a non-obstructive meniscal tear, and (2) to determine which patient factors direct surgeons towards APM and towards PT.

ELIGIBILITY:
In this survey the investigators invited orthopaedic surgeons and residents from both the Netherlands and Australia to complete a meniscus survey, including a random sample of patients from the Escape trial. The in-/exclusion criteria are listed below.

Inclusion Criteria:

* Patients between 45 and 70 years of age at presentation.
* A meniscal tear visualized on MRI. The meniscal tear can either be isolated or combined with a partial asymptomatic Anterior Cruciate Ligament (ACL) injury or an asymptomatic degenerative ACL shown on MRI with no abnormal clinical findings (a negative Lachman test and Pivot Shift).
* Mental Competence.
* Willingness to comply with follow up schedule.
* Written informed consent.

Exclusion Criteria:

* Knee locking or trauma leading to acute surgery.
* One of the following associated injuries on the index knee:
* A symptomatic partial ACL rupture or any total ACL rupture determined by clinical examination (positive Lachman test and/or positive Pivot Shift) and shown on MRI;
* A complete Posterior Cruciate Ligament (PCL) injury;
* Cartilage change down to bone; grade 4 of the Kellgren Lawrence Grading Scale for Osteoarthritis visualized on X-ray;
* An injury to the lateral/posterolateral ligament complex with significantly increased laxity.
* A history of knee surgery other than diagnostic arthroscopy on the index knee.
* Tumors on MRI suspected for a malignancy.
* Obese patients with Body Mass Index (BMI) > 35.
* ASA 4-5 patients which can severely interfere with rehabilitation.
* General disease that effects physical function or systemic medication/abuse of steroids (e.g., rheumatoid arthritis, psoriatic arthritis, systemic lupus erythematosus, gout, pseudogout)
* Any other medical condition or treatment interfering with the completion or assessment of the trial, e.g. contraindications to MRI or surgery.
* Drugs or alcohol abuse.

Ages: 45 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1. Orthopaedic surgeons and residents registered at the Dutch Orthopaedic Associations.
  2. A sample of orthopaedic surgeons from Australia
Sampling Method: Non-Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
The ability of orthopaedics surgeons to predict the outcome of treatment | 2 years
  In this survey, participants are provided with 20 cases and asked for their treatment of choice (APM or physical therapy). Subsequently, participants are asked for the expected outcome, which is change in knee function on the International Knee Documentation Committee 'Subjective Knee Form' (IKDC).
  These data are used to assess to what extend orthopaedic surgeons are capable of predicting the outcome of surgical and non-operative treatment of meniscal tears in a random sample of patients from the Escape trial.

SECONDARY OUTCOMES:
To assess which patient specific factors are found important by orthopaedic surgeons in choosing their treatment of first choice | 2 years
  In this survey, participants are asked to choose from a list of patient specific factors, which of these direct their treatment choice toward APM, and which towards non-operative treatment.
  These data are used to examine which patient specific factors are directing orthopaedic surgeons towards APM and towards PT. These factors will help future research focusing in creating patient specific profiles.

CONTACTS AND LOCATIONS:
Locations (1):
- Onze Lieve Vrouwe Gasthuis, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van de Graaf VA, Bloembergen CH MD, Willigenburg NW PhD, Noorduyn JCA MSc, Saris DB, Harris IA, Poolman RW; ESCAPE Research Group. Can even experienced orthopaedic surgeons predict who will benefit from surgery when patients present with degenerative meniscal tears? A survey of 194 orthopaedic surgeons who made 3880 predictions. Br J Sports Med. 2020 Mar;54(6):354-359. doi: 10.1136/bjsports-2019-100567. Epub 2019 Aug 1. PMID 31371339